CLINICAL TRIAL: NCT05419063
Title: Accessible Weight Loss: Examining the Feasibility of a Technology-Based Weight Loss Program for Adults With Low Vision
Brief Title: Accessible Weight Loss for Adults With Low Vision: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Towson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1535
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- weight loss program (Experimental): Participants will receive recommendations on how to decrease caloric intake, monitor their weight and track the related behaviors and progress. The weight loss program will provide asynchronous support (information, automated texting feedback, tailored emails) for adopting and maintaining lifestyle-based strategies for safe and effective weight loss.
  Interventions: Behavioral: weight loss strategies; Behavioral: text-based and email feedback

INTERVENTIONS:
Behavioral: weight loss strategies — Participants will receive recommendations on how to decrease caloric intake, monitor their weight and track the related behaviors and progress.
Behavioral: text-based and email feedback — Participants will receive weekly text-based feedback based on dietary strategy tracking and weight tracking. Participants will receive tailored email support and synchronous problem solving sessions as needed.

SUMMARY:
This study will examine the feasibility of an all-remote approach to enrollment in and implementation of an 8-week weight loss program for adults with low vision. The weight loss program will provide asynchronous support (information, automated texting feedback, tailored emails) for adopting and maintaining lifestyle-based strategies for safe and effective weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* English speaking
* BMI ≥ 25 and weight < 300lbs (weight limit due to scale limitations)
* Legally blind
* Have an email for personal use and ability to check and respond to email daily
* Have a smart phone with texting for personal use
* Sufficient internet plan for daily email checking
* Sufficient phone plan for 12 or more texts per week
* Ability to send and receive emails and text messages
* Ability to join a zoom call on a personal phone, tablet, or computer
* Ability to complete Qualtrics surveys
* Willing to lose weight through recommended dietary changes, weight tracking and physical activity
* Interest in one of the specific dietary strategies supported by the text messaging platform
* Willing to use the study scale with cellular technology to report weights
* Willing to join an 8-week weight loss program and interested in losing weight
* Completion of screening, enrollment and baseline data collection

Exclusion Criteria:

* Lost 5% of body weight in the last 6 months
* Currently participating in a weight loss program or another weight loss study
* Previously diagnosed eating disorder, or treatment for an eating disorder
* Pregnant, nursing, or planned pregnancy in the next 6 months
* Planned weight loss surgery or procedure in the next 6 months
* Currently using medication for weight loss (prescribed or over the counter)
* History of cardiovascular events
* History of type 1 or type 2 diabetes
* Prescribed medication that might promote weight change such as lithium, steroids, or antipsychotics
* Medical contraindicate to weight loss (e.g., end-stage renal disease, cancer diagnosis with active/planned treatment)
* Psychiatric hospitalization in the past 12 months
* Investigator discretion for safety or to ensure appropriate treatment of study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Usability and helpfulness of program components at week 4 | week 4
  Using descriptive statistics, examine 5-point Likert scale responses for the usability (0 = not at all easy to use; 4= extremely easy to use) and helpfulness (0 = not at all helpful; 4= extremely helpful) of specific program components at week 4.

SECONDARY OUTCOMES:
Usability and helpfulness of program components at week 8 | week 8
  Using descriptive statistics, examine 5-point Likert scale responses for the usability (0 = not at all easy to use; 4= extremely easy to use) and helpfulness (0 = not at all helpful; 4= extremely helpful) of specific program components at week 8.
Program engagement at weeks 4 and 8 | week 4 and 8
  Examine the percentage of weeks with at least one study weight and the percentage of days with responses to dietary tracking at weeks 4 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Jerome, Principal Investigator — Towson University
Locations (1):
- Towson University, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Depuy J, Molina-Morales J, Conover AJ, Jerome GJ. Accessible weight loss program for adults who are legally blind: A pilot study. Disabil Health J. 2023 Oct;16(4):101502. doi: 10.1016/j.dhjo.2023.101502. Epub 2023 Jul 4. PMID 37482499